CLINICAL TRIAL: NCT04293718
Title: Acquired Chronic Erosive Gingivitis: Clinical Relevance of Papillary Gingival Biopsy. Retrospective Bicentric Study of 148 Samples and Systematic Review of the Literature
Brief Title: Acquired Chronic Erosive Gingivitis: Clinical Relevance of Papillary Gingival Biopsy
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: ODONT_APHP_HMN2019
Record Dates: First submitted 2020-02-20; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-01

CONDITIONS: Gingival Diseases; Gingivitis; Autoimmune Diseases; Oral Lichen Planus
Keywords: Erosive gingivitis; Biopsy; Desquamative gingivitis; Gingival disease; Oral lichen planus; Mucous membrane pemphigoid benign; Pemphigus vulgaris
MeSH Terms: conditions — Gingival Diseases; Gingivitis; Autoimmune Diseases; Lichen Planus, Oral; Pemphigoid, Benign Mucous Membrane; Pemphigus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Gingival biopsies were performed. At least one biopsy per patient was intended for anatomopathological examination; a second biopsy was required for direct immunofluorescence (DIF), for generalized, particularly severe erosive gingivitis, and/or in the presence of pseudomembranes, gingival or oral blisters suggesting the existence of an autoimmune bullous disease with gingival expression. This second biopsy was performed either in the wake of the first or in second line after reading the first anatomopathological examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute erosive gingivitis: Patients presenting acute erosive gingivitis, isolated or predominant compared to other oral lesions, which required at least one papillary gingival biopsy for diagnostic purposes. Patients were included in the study regardless of age and general health.
  Interventions: Other: papillary gum biopsies

INTERVENTIONS:
Other: papillary gum biopsies — 1 or 2 papillary gum biopsies were performed simultaneously, 1 for histological examination and 1 for immunohistochemistry

SUMMARY:
Chronic erosive gingivitis is a syndrome (CEGS) that combines severe gingival inflammation and gingival erosion. The term "desquamative gingivitis" is often used in the literature to define chronic erosive gingivitis. However, this definition is inappropriate because the pathophysiological process at the origin of this gingival disease does not induce a desquamation but rather a loss of gingival substance, namely erosion, concerned wholly or in part of the gingival epithelium. In most clinical situations, chronic erosive gingivitis is an oral manifestation of a general disease with immune dysfunction. The most frequently described diseases are gingival lichen and autoimmune bullous diseases (AIBD). In 2018, as part of a monocentric study, we were the first to detail an original papillary gingival biopsy protocol, non-iatrogenic, perfectly suited to the anatomopathological examinations necessary for the diagnosis of AIBD gingival expression. The CEGS early detection by odontologists avoid delayed diagnosis and allows patients to be referred to the closest AIBD reference center.

Hypothesis/Objective A bicentric study was conducted, to evaluate the clinical relevance of this protocol, including the differential diagnosis of the CEGS. Research was supplemented by carrying out a systematic review of the literature to compare the contributive capacity diagnostic of the papillary biopsy technique with other gingival sample methods (attached gingival tissue, mucosa).

Method A retrospective bicentric observational study was conducted from October 2011 to July 2019, in two departments of oral medicine of two public hospitals in Paris (University Hospital - Bretonneau in Paris and Henri Mondor in Créteil; France). These two departments are specialized in the diagnosis and management of oral pathology; that of the Henri Mondor hospital is an AIBD reference center.

The literature review was developed in accordance with PRISMA recommendations. It was conducted on Pubmed - MEDLINE and Cochrane Oral Health Group and included all existing publications from 1935 until August 2019. A manual search of publications from the unpublished literature was also conducted.

ELIGIBILITY:
Inclusion Criteria:

• Patients referred on an outpatient basis by the physician or the dental surgeon, suffering from an acute erosive gingivitis, regardless of age and general health.

Exclusion Criteria:

• Patients referred on an outpatient basis by the physician or the dental surgeon, with a histological examination and immunofluorescence (DIF) already done previously, and patient under corticosteroid therapy which is skewing the immunofluorescence (DIF) data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over the study period we were able to study 101 files, but the investigator's final sample of patients included 100 adults. In first-line, 2 papillary gum biopsies were performed simultaneously for 48 of them (48%), 1 for histological examination and 1 for immunohistochemistry. For 47 other patients (47%) only 1 biopsy was performed for histological examination and for the remaining 5 patients (5%) only 1 biopsy for immunofluorescence (DIF).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
contributive capacity diagnostic of the papillary biopsy technique | One week after biopsy has been performed
  Diagnosis of certainty of diseases, whose clinical features are the CEGS, have been made by comparing clinical data with histological criteria commonly accepted by the international community
  One week after the biopsy has been performed, we can establish the:
  * number of contributive results of first-line biopsies performed for conventional histological analysis showing the:
    * presence or absence of the epithelium,
    * presence or absence of the intra-epithelial or the subepithelial cleavage,
    * characteristic of the inflammatory infiltrate, especially the presence and the number of lymphocytes.
  * number of contributive results of biopsies performed for direct immunofluorescence showing:
    * immune deposits or not, in a linear staining pattern at the chorio-epithelial junction.
    * immune deposits or not, in an intercellular staining pattern in the epidermis.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Position paper: oral features of mucocutaneous disorders. J Periodontol. 2003 Oct;74(10):1545-56. doi: 10.1902/jop.2003.74.10.1545. PMID 14653403
- [Background] Cheng YS, Gould A, Kurago Z, Fantasia J, Muller S. Diagnosis of oral lichen planus: a position paper of the American Academy of Oral and Maxillofacial Pathology. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Sep;122(3):332-54. doi: 10.1016/j.oooo.2016.05.004. Epub 2016 Jul 9. PMID 27401683
- [Background] Dridi SM, Bellakhdar F, Ortonne N, Bayet K, Ingen-Housz-Oro S, Gaultier F. [Autoimmune bullous diseases with gingival expression: A proposed non-iatrogenic gingival biopsy technique]. Ann Dermatol Venereol. 2018 Oct;145(10):572-577. doi: 10.1016/j.annder.2018.06.005. Epub 2018 Aug 22. French. PMID 30143321
- [Background] Lo Russo L, Fedele S, Guiglia R, Ciavarella D, Lo Muzio L, Gallo P, Di Liberto C, Campisi G. Diagnostic pathways and clinical significance of desquamative gingivitis. J Periodontol. 2008 Jan;79(1):4-24. doi: 10.1902/jop.2008.070231. PMID 18166088
- [Background] Rinaggio J, Crossland DM, Zeid MY. A determination of the range of oral conditions submitted for microscopic and direct immunofluorescence analysis. J Periodontol. 2007 Oct;78(10):1904-10. doi: 10.1902/jop.2007.070095. PMID 18062112
- [Background] van der Meij EH, van der Waal I. Lack of clinicopathologic correlation in the diagnosis of oral lichen planus based on the presently available diagnostic criteria and suggestions for modifications. J Oral Pathol Med. 2003 Oct;32(9):507-12. doi: 10.1034/j.1600-0714.2003.00125.x. PMID 12969224
- [Derived] Gaultier F, Ejeil AL, Jungo S, Ingen-Housz-Oro S, de Clatigny FLP, Bruno G, Pirnay P, Bellakhdar F, Dridi SM. Clinical relevance of interdental papilla biopsy in chronic erosive gingivitis (desquamative gingivitis): retrospective bicentric study of 148 specimens. BMC Oral Health. 2021 Sep 17;21(1):452. doi: 10.1186/s12903-021-01820-9. PMID 34535102